CLINICAL TRIAL: NCT04111380
Title: Efficacy and Safety of Nab-Paclitaxel Combined With Cisplatin in Second or Later-Line Treatment in Advanced Biliary Tract Cancers: a Prospective, Open Label, Single-arm Phase II Trial
Brief Title: Efficacy and Safety Study of Nab-Paclitaxel Combined With Cisplatin in Second or Later-Line Treatment in Advanced Biliary Tract Cancers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jianwei Zhou
Record Dates: First submitted 2019-09-29; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Advanced Biliary Tract Cancers
MeSH Terms: interventions — Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel and Cisplatin (Experimental): cisplatin and nab-paclitaxel: Nab-paclitaxel, 130mg/m2, d1,d8, Cisplatin, 20mg/m2, d1-3 ,3week, 4-6 cycles.
  Interventions: Drug: cisplatin and nab-paclitaxel

INTERVENTIONS:
Drug: cisplatin and nab-paclitaxel — Nab-paclitaxel, 130mg/m2, d1,d8, Cisplatin, 20mg/m2, d1-3 ,3week, 4-6 cycles.

SUMMARY:
To verify the role of nab-paclitaxel in second or later-line treatment in advanced biliary tract cancers, the investigators designed a prospective, exploratory, single arm,single center phase II trial, to investigate the efficacy and safety of nab-paclitaxel combined with cisplatin as second or later-line treatment in advanced biliary tract cancers.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 18 to 75 years
* Radiographically, histologically or/and cytologically diagnosed intrahepatic cholangiocarcinoma, extrahepatic cholangiocarcinoma, or gallbladder cancer.
* Received at least one first-line systemic treatment for advanced or metastatic diseases and failed, with imaging evidence of disease progression.
* ECOG performance status 0-1
* According to the RECIST1.1 standard, at least one measurable objective lesion should be judged.
* Expected survival more than 12 weeks
* The laboratory test meet the following requirements:

Bone marrow function: neutrophils ≥ 1.5×10(9)/L, platelets ≥ 100×10(9)/L, hemoglobin ≥ 90 g/L Liver function：Total bilirubin ≤ 1.5x ULN；AST and ALT) ≤ 2.5x ULN Renal function：Cr ≤ 1.5x ULN，Ccr ≥ 45 ml/min Coagulation function：INR≤1.5×ULN, PT≤1.5ULN, APTT within the normal range

* Not concomitant with other uncontrollable benign disease before the recruitment(e.g. the infection in the kidney, lung and liver).
* During the non-lactation period, contraceptive measures should be taken in patients of child-bearing age during this trial. The test ofβ- HCG was negative.
* The patient has good compliance with the planned treatment, understands the research process of the study and signs a written informed consent form

Exclusion Criteria:

* With Chemotherapy contraindication, known to be allergic, highly sensitive or intolerable to research-related drugs or excipient.
* Pregnant or lactating women.
* Refuse or fail to sign informed consent to participate in the trial
* Grade 2 or above peripheral neuropathy or hemorrhage according to NCI CTCAE 4.03
* Combined with severe cardiovascular disease, including hypertension that cannot be controlled by medical treatment(BP≥160/95mmHg), unstable angina, a history of myocardial infarction in the past 6 months,Congestive heart failure>NYHA grade II, severe arrhythmia, pericardial effusion, etc.
* Patients with severe systemic infections or other serious diseases.
* Combined with other primary tumors
* Patients not suitable for the group according to the judgement of the researcher, with mental disease.
* Patients with symptomatic central nervous system (CNS) metastases who require radiotherapy, surgery or sustained corticosteroid use, and untreated brain metastases that cause any symptoms
* Prior exposure to nab-paclitaxel
* The investigator determined that unable to complete the study due to medical, social, or psychological reasons or were unable to sign valid informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate [ORR] | 2 years

SECONDARY OUTCOMES:
Progression Free Survival [PFS] | 2 years
Overall survival [OS] | 2 years
Disease Control Rate [DCR] | 2 years
adverse events | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology , Henan Provincial People's Hospital, People's Hospital of Zhengzhou University, People's Hospital of Henan University, Zhengzhou, Henan, China